CLINICAL TRIAL: NCT05234099
Title: Evaluation of the Sensitivity and Reproducibility of 18F-fluorodeoxyglucose Positron Emission Tomography Coupled With Magnetic Resonance Imaging for the Assessment of Respiratory Muscle Activity and Relationships With Multiparametric Respiratory Muscle Ultrasound
Brief Title: Sensitivity and Reproducibility of 18F-fluorodeoxyglucose Positron Emission Tomography for Assessment of Respiratory Muscle Activity
Acronym: ResPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ResPET
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Muscle
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control subjects (Experimental): Visit 1 (V1) (Duration: 2.5h)
  * Information, verification of inclusion and exclusion criteria, information note.
  * Consent form.
  * Location of the diaphragm and parasternal intercostal muscle using ultrasound.
  * Measurements at rest (mouth pressures, sEMG, ultrasound imaging).
  * Injection of 3 MBq/kg of 18F-FDG.
  * 1h resting period.
  * 18F-FDG PET-MRI scan.
  Visit 2 (V2) 3-10 days after V1 (Duration: 3h)
  * Location of the diaphragm and parasternal intercostal muscle.
  * Measurements at rest (mouth pressures, sEMG, ultrasound imaging)
  * Magnetic stimulation of the phrenic nerves
  * Ventilation against inspiratory loading
  * Magnetic stimulation of the phrenic nerves
  * Injection of 3 MBq/kg of 18F-FDG
  * 1h resting period
  * 18F-FDG PET-MRI scan
  Visit 3 (V3) 3-10 days after V2 (Duration: 3h)
  - Identical to visit 2
  Interventions: Diagnostic Test: 18F-FDG Positron emission tomography - MRI; Diagnostic Test: Multiparametric ultrasound imaging; Diagnostic Test: Surface electromyography; Diagnostic Test: Transdiaphragmatic preasure measurmement; Diagnostic Test: Magnetic stimulation of the phrenic nerves; Diagnostic Test: Ventilation against inspiratory loading

INTERVENTIONS:
Diagnostic Test: 18F-FDG Positron emission tomography - MRI — All the examinations will be performed in the supine position on the same integrated 3T PET-MRI scanner
Diagnostic Test: Multiparametric ultrasound imaging — Acquisitions of respiratory muscles (diaphragm, intercostal muscles) will be performed using two 6 MHz central frequency linear transducer (SL 10-2) driven by two identical ultrafast ultrasound devices.
Diagnostic Test: Surface electromyography — sEMG recordings will be performed in the left side on the sternocleidomastoid muscle, the intercostal parasternal muscle, and the external oblique muscle using pairs of 20-mm-diameter silver chloride surface electrodes.
  Other Names: sEMG
Diagnostic Test: Transdiaphragmatic preasure measurmement — Esophageal and gastric pressures will be measured using 8-cm balloon-catheters.
  Other Names: Internal respiratory pressures measurements
Diagnostic Test: Magnetic stimulation of the phrenic nerves — In order to quantify the contractile fatigue in diaphragm induced by the ventilatory task (described below), we will use bilateral anterior magnetic stimulation of the phrenic nerves using two Magstim 200 stimulator.
Diagnostic Test: Ventilation against inspiratory loading — A POWERbreathe KH2 device (POWERbreathe International Ltd) will be connected on the inspiratory side of the two-way valve. Level of inspiratory loading will be randomized in order to produce different amounts of muscle work in each subject.

SUMMARY:
The assessment of respiratory muscle function is critical within both clinical and research settings. Tools for the assessment of respiratory muscle function are especially useful in diagnosing, phenotyping, understanding pathophysiology, and assessing treatment responses in patients with respiratory symptoms, including critically hill patients and patients with respiratory and/or neuromuscular diseases. Respiratory muscle function is most commonly assessed using flow (i.e. spirometry) and pressure measurements during spontaneous ventilation, voluntary respiratory efforts, or artificially evoked responses using magnetic or electrical stimulation. Some of these approaches may be limited within patients suffering from neuromuscular diseases. The study hypothesis is the 18F-FDG PET technology, heavily used for clinical oncology purposes (diagnostic, staging, response to treatment, prognosis), could be an interesting alternative to invasive measurement of the respiratory muscle activity. In addition, it may contribute to further validate metrics based on multiparametric ultrasound imaging.

DETAILED DESCRIPTION:
The assessment of respiratory muscle function is critical within both clinical and research settings. Tools for the assessment of respiratory muscle function are especially useful in diagnosing, phenotyping, understanding pathophysiology, and assessing treatment responses in patients with respiratory symptoms, including critically hill patients and patients with respiratory and/or neuromuscular diseases. Respiratory muscle function is most commonly assessed using flow (i.e. spirometry) and pressure measurements during spontaneous ventilation, voluntary respiratory efforts, or artificially evoked responses using magnetic or electrical stimulation. Some of these approaches may be limited, for instance, when facial muscle weakness occurs and/or when glottis function is compromised, for example in patients with bulbar amyotrophic lateral sclerosis or myopathies. Consequently, widely used respiratory measures can be poor predictors of respiratory muscle alterations and this may contribute to affect clinical decisions such as the time when non-invasive ventilation should be initiated within the disease continuum.

Positron emission tomography (PET) is a nuclear medicine procedure based on the measurement of positron emission from radiolabeled tracer molecules. These radiotracers allow biologic processes to be measured and whole-body images to be obtained which demonstrates sites of radiotracer accumulation. Fluorodeoxyglucose (18F-FDG) is a radiolabeled glucose molecule and is the most common radiotracer used in clinical practice. 18F-FDG PET is most frequently coupled with computed tomography but may also be coupled with magnetic resonance imaging (18F-FDG PET-MRI). 18F-FDG PET is heavily used for clinical oncology purposes (diagnostic, staging, response to treatment, prognosis). 18F-FDG PET also finds applications in other fields for detecting infections and inflammatory processes. 18F-FDG may also be used in muscles that are major user of glucose. 18F-FDG PET offers the opportunity to assess the patterns and work amount of multiple muscles simultaneously, providing a global view of the muscles involved in the realization of a motor task, as previously demonstrated in shoulder muscles.

Ultrasound imaging (US) is attracting a growing interest for the assessment of respiratory muscle function, as it allows bedside and non-invasive assessments. Recently, new US techniques such as shear wave elastography (SWE) have shown promises for the assessment of respiratory muscle work. However, the ability of variables derived from respiratory muscle US to reflect increased muscle work remains unclear. Hence, building evidences supporting non-invasive US biomarkers for respiratory muscle function is necessary.

18F-FDG PET offers a unique opportunity to investigate patterns and work amount of the respiratory muscles. In a resting state, 18F-FDG uptake in the respiratory muscle is known to be small. However, and to the best of our knowledge, 18F-FDG uptake of the respiratory muscles at rest in healthy subjects has never been specifically reported. It is unclear whether 18F-FDG PET may be used to monitor changes in respiratory muscle activity within the disease continuum or in response to an intervention such as the initiation of non-invasive ventilation. The reproducibility of increase 18F-FDG uptake of the respiratory muscles induced remains to be assessed and is a prerequisite to determine its sensitivity to change. Moreover, the relationship between increase 18F-FDG uptake and respiratory muscle work as assessed using other methods (e.g. flow and pressure measurements, surface electromyography (sEMG)) and variables derived from multiparametric US remains to be determined. Since MRI does not use ionizing radiations, and because of very higher soft-tissue contrast capabilities, combining PET to MRI instead of CT is of better relevance for our PET muscular analyses purpose.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yo
* Non-smoker
* Signed informed consent
* Affiliate or beneficiary of a social security scheme

Non-Inclusion Criteria:

* Pregnant or breastfeeding women
* Respiratory, cardiovascular, metabolic, neuromuscular pathologies
* Claustrophobia
* Belonephobia
* Latex allergy
* Persons subject to a legal protection measure or unable to express their consent
* Contraindications to MRI (claustrophobia, metal implants)
* Inability to participate in the study
* Inability to comply with protocol requirements

Exclusion Criteria:

* Blood sugar> 1.8 g / L (V1, V2, V3)
* Impossibility of inserting the esophageal and / or gastric tubes (V2, V3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Correlation between multiparametric ultrasound and 18F-FDG PET-MRI during respiratory muscle activity measurement | Through study completion, on average 3 weeks
  Existence of a significant correlation between the variables derived from the multiparametric ultrasound and the work of the respiratory muscles induced by the ventilatory spot assessed by 18F-FDG PET-MRI

SECONDARY OUTCOMES:
Significant correlation between measurements of respiratory muscle activity assessed by pressure measurements and increased respiratory muscle work induced by the ventilation against inspiratory loading as assessed by 18F-FDG PET-MRI | Through study completion, on average 3 weeks
  Existence of a significant correlation between measurements of respiratory muscle activity assessed by pressure measurements (esophageal pressure, gastric pressure, transdiaphragmatic pressure) and increased respiratory muscle work induced by the ventilation against inspiratory loading as assessed by 18F-FDG PET-MRI
Significant correlation between measures of respiratory muscle activity assessed by sEMG and respiratory muscle work induced by the ventilation against inspiratory loading as assessed by 18F-FDG PET-MRI | Through study completion, on average 3 weeks
  Existence of a significant correlation between measures of respiratory muscle activity assessed by sEMG and respiratory muscle work induced by the ventilation against inspiratory loading as assessed by 18F-FDG PET-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Damien Bachasson, PhD, Principal Investigator — Institute of Myology
Locations (2):
- France (2):
  - Service hospitalier Fréderic Joliot, Orsay
  - Association Institut de Myologie, Paris